CLINICAL TRIAL: NCT03352505
Title: Associations Between the Cardiovascular Risk Markers and Neuroplasticity in Sedentary or Physically Active Spinal Cord Injured Subjects of the Wheelchair Dancer Study
Brief Title: Cardiovascular Risk Markers in Spinal Cord Injured Subjects of the Wheelchair Dancer Study
Status: Completed | Type: Observational
Sponsor: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Prof. Josef Niebauer M.D., Ph.D., MBA, Prof. Josef Niebauer, M.D., Ph.D, MBA, Paracelsus Medical University
Other Study IDs: UISM-12
Record Dates: First submitted 2017-11-16; First posted 2017-11-24 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: SCI - Spinal Cord Injury; Cardiovascular Risk Factor
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control: healthy walking control participants
- wheelchair dancer: wheelchair users, who are performing wheelchair dancing
- wheelchair marathon participants: wheelchair users, who are participants in wheelchair/ handbike Marathon competitions
- sedentary wheelchair patients: wheelchair users, who conduct exercise bouts less than 2 times per month

SUMMARY:
The present study will analyze if exercise is able to elicit the well-known anti-atherogenic effects in patients with SCI. This will be evaluated by measuring vascular parameters such as endothelial and inflammatory blood markers, echocardiography of the heart and peripheral vessels, as well as blood pressure and arterial stiffness, in subjects performing either wheelchair dancing, wheelchair marathon or no sports. Further, it will be investigated, whether there is an association between neuroplasticity and cardiovascular health, as measured by electroencephalography (EEG), transcranial magnetic stimulation (TMS) and blood levels of the brain-derived neurotrophic factor (BDNF).

We hypothesize that the cardiovascular, physical and psychological benefits of wheelchair dancing and/or wheelchair marathon parallel improved neuroplasticity in SCI-patients

ELIGIBILITY:
Inclusion Criteria:

wheelchair users independent of the cause of the walking impairment, preferably with spinal cord injury.

Exclusion Criteria:

metallic implanters, additional neurologic pathologies, pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy participants, wheelchair users
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
comparison of cardiovascular risk factors between different study groups | October 2017- June 2018
  measurement for arterial stiffness parameters, via pulse wave analysis. Comparison between healthy individuals and patients using wheelchairs (three different groups).
Evaluation of echocardiography results between different study groups | October 2017- June 2018
  Evaluation of echocardiography comparing healthy individuals and patients using wheelchairs (three different groups).

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Department of Neurology, Christian Doppler Klinik, Paracelsus Medical University Salzburg, Salzburg
  - Department of Sports Medicine, Prevention and Rehabilitation Paracelsus Medical University, Salzburg